CLINICAL TRIAL: NCT06609200
Title: Electro-acupuncture for the Obese Patient with Insulin Resistance: a Randomized Sham-controlled Clinical Trial
Brief Title: Electro-Acupuncture for Obese Patients with Insulin Resistance
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanyang Technological University (Other)
Responsible Party: Principal Investigator, Linda Zhong, Assoc prof, Nanyang Technological University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-2024-165
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Obesity; Insulin Resistance
Keywords: electroacupuncture; obesity; insulin resistance
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Each patient will be scheduled for 16 treatment sessions, each lasting 30 minutes, twice a week over 8 weeks.
Who Masked: Participant, Outcomes Assessor
Masking Description: After a participant's eligibility is confirmed, a randomization number that corresponds to the group allocation will be provided to the acupuncturist. The clinical assessor and participants will be blinded to the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Electroacupuncture group (Experimental): The WHO Standardized Acupuncture Points Location [2] will be used to identify the location of these acupoints, Tianshu(ST-25), Daheng(SP-15), Daimai(GB-24), Qihai(CV-6), Zhongwan(CV-12), Zusanli (ST-36), Fenlong(ST-40), and Sanyinjiao(SP-6). After sterilizing the skin, sterile adhesive pads will be pasted on acupoints first, and then needles of size 0.30*75 mm will be inserted into the acupoints to a depth of 50 mm outward and upward slightly. Needles will be lifted, thrust, and twirled evenly 3 times to achieve "de-qi". Paired electrodes of the EA apparatus will be attached transversely to the acupoint respectively with a continuous wave of 50 Hz and a current intensity of 1-5 mA (preferably with the skin around the acupoints shivering mildly without pain) for 30 min. Patients will be treated with electroacupuncture 2 sessions per week over 8 consecutive weeks, 16 sessions for each patient.
  Interventions: Device: Acupuncture needles
- Sham acupuncture group (Sham Comparator): The sham electro-acupuncture group (SEA) penetrates acupuncture on non-acupuncture points (1 cm away from the acupuncture point and meridian). The same type of acupuncture needles will be used for SEA with the exact skin sterilization method. All acupuncture points will be needled perpendicularly with a guide tube. Insertion depth will be approximately 50 mm, depending on the location of individual points. Each point will be connected to a sham electro-stimulator (showing a continuous wave at a frequency of 30 Hz but without actual stimulation). All needles will be removed after 30 min of needle retention. Patients will be treated with sham electroacupuncture 2 sessions per week over 8 consecutive weeks, 16 sessions for each patient in total.
  Interventions: Device: Acupuncture needles

INTERVENTIONS:
Device: Acupuncture needles — The acupuncture needles and related equipment will have already received approval for routine Traditional Chinese Medicine (TCM) clinical practice in Singapore.

SUMMARY:
This clinical trial aims to evaluate the efficacy and safety of electro-acupuncture for obese patients with insulin resistance. 60 participants will be randomized and allocated to either the electro-acupuncture arm or the sham acupuncture arm.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 21 and 65 years old
* BMI ≥ 25 kg/m2
* HOMA-IR ≥ 2.14, (HOMA-IR = fasting insulin (ųU/mL)* fasting glucose (mmol/L)/22.5)
* Not receiving any other weight control measures or any medical and/or drug history in the last 3 months

Exclusion Criteria:

* Diabetes mellitus
* Treating with drugs that may affect insulin sensitivity
* Changes 10% of usual body weight in the previous 6 months weight
* Endocrine diseases, including thyroid disorder, pituitary disorder, sex gland disorder, etc.
* Heart diseases, including arrhythmia, heart failure, and myocardial infarction, participants with pacemakers
* Allergy and immunology diseases
* Bleeding tendency
* Pregnant or lactating women
* Impaired hepatic or renal function
* Stroke or unable to exercise

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-10 (Estimated); Primary Completion 2026-04-09 (Estimated); Study Completion 2026-10-09 (Estimated)

PRIMARY OUTCOMES:
HOMA-IR | From enrollment to the end of follow up at 16 weeks
  HOMA-IR = fasting insulin (ųU/mL)* fasting glucose (mmol/L)/22.5

SECONDARY OUTCOMES:
Body Mass Index (BMI) | From enrollment to the end of follow up at 16 weeks
  BMI = kg/m2
Waist-to-hip ratio | From enrollment to the end of follow up at 16 weeks
  The waist-hip ratio or waist-to-hip ratio (WHR) is the dimensionless ratio of the circumference of the waist to that of the hips.

IPD SHARING:
Plan to Share IPD: Yes
IPD sharing will be available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available within 7 years after completion of the clinical trial.
Access Criteria: Individual participant data (IPD) will be made available to qualified researchers upon request. To access the data, researchers must submit a formal request, which will be reviewed and approved by the data-sharing committee. Data access will be granted for research purposes only and will require adherence to data use agreements and ethics guidelines.